CLINICAL TRIAL: NCT06162416
Title: Non-opioid Anesthesia in Bariatric Surgery
Acronym: BARIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7645
Record Dates: First submitted 2022-11-08; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Severe Obesity
Keywords: Bariatric surgery; Opioid-free anesthesia; Non-opioid anesthesia; Severe obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Opioid-free anesthesia is a new approach to anesthesia, described and used for many years. If it represents many advantages by reducing the side effects of morphine, its precise place in current practice and in terms of postoperative rehabilitation remains to be determined. Studies are not yet numerous enough to affirm a real benefit.

Obese patients are potentially able to benefit from the reduction in the use of morphine during surgery, in terms of quality of postoperative analgesia, side effects (respiratory depression, ileus, somnolence) and early rehabilitation.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥ 18 years old),
* who have undergone bariatric surgery at the HUS between January 01, 2017 and December 31, 2019
* Subject who has not expressed his or her opposition, after information, to the reuse of his or her data for the purpose of this research

Exclusion Criteria:

* Subject who has expressed his/her opposition to participate in the study
* Subjects under guardianship, curatorship or legal protection, pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years old) who have undergone bariatric surgery at the HUS between January 01, 2017 and December 31, 2019
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose of morphine used intraoperatively | Intraoperative (during the operation)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France